CLINICAL TRIAL: NCT07298772
Title: A Phase Ib/II, Multicenter, Open-Label Study of Safety, Tolerability and Efficacy of SHR-4375 Injection in Combination With Other Antitumor Therapies in Patients With Advanced Solid Tumors
Brief Title: A Study of SHR-4375 Injection in Combination With Other Antitumor Therapies in Patients With Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4375-201
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Bevacizumab; Fluorouracil; Leucovorin; Paclitaxel; Injections; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental)
  Interventions: Drug: SHR-4375 Injection; Drug: Paclitaxel for injection
- Arm B (Experimental)
  Interventions: Drug: SHR-4375 Injection; Drug: Bevacizumab Injection; Drug: Fluorouracil injection; Drug: Calcium Folinate Injection
- Arm C (Experimental)
  Interventions: Drug: SHR-4375 Injection; Drug: Bevacizumab Injection; Drug: Fluorouracil injection; Drug: Calcium Folinate Injection; Drug: Oxaliplatin injection

INTERVENTIONS:
Drug: SHR-4375 Injection — SHR-4375 injection.
Drug: Bevacizumab Injection — Bevacizumab injection.
  Arms: Arm B; Arm C
Drug: Fluorouracil injection — Fluorouracil injection.
  Arms: Arm B; Arm C
Drug: Calcium Folinate Injection — Calcium Folinate injection.
  Arms: Arm B; Arm C
Drug: Paclitaxel for injection — Paclitaxel for injection.
  Arms: Arm A
Drug: Oxaliplatin injection — Oxaliplatin injection.
  Arms: Arm C

SUMMARY:
This is an open label, multi-center, Phase Ib/II study to evaluate the safety, tolerability and efficacy of SHR-4375 injection in combination with other antitumor therapies in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18-75 years older, no gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
4. With a life expectancy ≥ 12 weeks.
5. Patients with advanced solid tumors confirmed by cytology or histology who have failed or are intolerant to standard treatment and have no standard treatment.
6. Be able to provide fresh or archived tumour tissue.
7. At least one measurable lesion according to RECIST v1.1.
8. Adequate bone marrow and organ function.
9. Contraception is required during clinical trials, and pregnancy tests must be negative for women of childbearing age within 7 days before the first dose.

Exclusion Criteria:

1. There are components of neuroendocrine carcinoma or sarcoma in the histopathological type.
2. Had received chemotherapy, immunotherapy, targeted therapy, anti-tumor traditional Chinese medicine or other clinical research drugs within 4 weeks prior to the first administration of the study; Palliative radiotherapy was received within 2 weeks before the first administration.
3. Live attenuated vaccines are used within a certain period of time before the first medication as stipulated in the plan, or it is expected that such vaccines will be needed during the treatment period.
4. Having undergone major surgeries other than diagnosis or biopsy within 28 days prior to the first administration.
5. Previously received antibody-drug conjugate therapy containing topoisomerase I inhibitors.
6. Currently participating in other clinical studies or taking medication for the first time less than 4 weeks after the end of the previous clinical study.
7. Suffering from other active malignant tumors within 3 years or at the same time.
8. Symptomatic or active central nervous system tumor metastasis.
9. Accompanied by uncontrolled tumor related pain.
10. Subjects who have experienced severe infections within 30 days prior to their first medication use.
11. History of interstitial pneumonia/non infectious pneumonia requiring hormone therapy in the past.
12. AE caused by previous anti-tumor treatment has not recovered to CTCAE v5.0 level evaluation ≤ 1.
13. Active hepatitis B or active hepatitis C.
14. Clinically significant bleeding symptoms or significant bleeding tendency occurred within 1 month before the first medication.
15. Moderate and severe ascites with clinical symptoms; Uncontrolled or moderate to excessive pleural effusion and pericardial effusion.
16. Uncontrollable mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse, and criminal detention.
17. Per the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT). | 3 weeks.
Recommended phase II dose (RP2D). | From screening period up to study completion, an average of 1 year.
Adverse events (AEs). | From screening period up to study completion, an average of 1 year.
Objective response rate (ORR). | From screening period up to study completion, an average of 1 year.

SECONDARY OUTCOMES:
Disease control rate (DCR) | From screening period up to study completion, an average of 1 year.
Duration of response (DoR) | From screening period up to study completion, an average of 1 year.
Progression-free survival (PFS) | From screening period up to study completion, an average of 1 year.
Drug Resistant Antibody (ADA) to SHR-4375 | From screening period up to study completion, an average of 1 year.
  Immunogenicity: The number of subjects with ADA to SHR-4375, incidence, time of occurrence, duration, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided